CLINICAL TRIAL: NCT05573373
Title: Double Arm Single Center Clinical Trial of Pamiparib (BGB-290) for EGFR TKIs Resistant Non-small Cell Lung Cance
Brief Title: Pamiparib (BGB-290) Was Used in EGFR-TkIs Resistant Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 136266
Record Dates: First submitted 2022-09-22; First posted 2022-10-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; EGF-R Positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pamiparib; Poly A; Adenosine Diphosphate Ribose; Antineoplastic Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pamilarib in combination with Chemotherapy Drugs (Experimental): The specific chemotherapy regimen was formulated by the investigator. The dosage of chemotherapy drugs is selected according to the drug use guidelines. Combination medication, the initial dose is 40mg each time (2 capsules), 2 times a day, the total daily dose is 80mg. Can be taken with a meal or on an empty stomach. If the patient misses a dose, no additional dose should be taken, and the next prescribed dose should be taken normally at the planned time. Continue the treatment until the disease progresses or unacceptable adverse reactions occur, and the dose is adjusted.
  Interventions: Drug: Parimparib; Drug: Chemotherapy drug
- Pamiparib in combination with Targeted Therapy Drugs (Experimental): The specific targeted therapy plan is formulated by the investigator. The dosage of targeted therapeutic drugs is selected according to the drug use guidelines. Combination medication, the initial dose is 40mg each time (2 capsules), 2 times a day, the total daily dose is 80mg. Can be taken with a meal or on an empty stomach. If the patient misses a dose, no additional dose should be taken, and the next prescribed dose should be taken normally at the planned time. Continue the treatment until the disease progresses or unacceptable adverse reactions occur, and the dose is adjusted.
  Interventions: Drug: Parimparib; Drug: Targeted Therapy Agent

INTERVENTIONS:
Drug: Parimparib — The dosage and protocol of the drug were carried out according to the description.
  Other Names: BGB-290; Poly (ADP-ribose) polymerase (PARP) inhibitor
Drug: Chemotherapy drug — The dosage and protocol of the drug were carried out according to the description.
  Other Names: Chemotherapy Drug, Cancer
  Arms: Pamilarib in combination with Chemotherapy Drugs
Drug: Targeted Therapy Agent — The dosage and protocol of the drug were carried out according to the description.
  Other Names: Targeted drug
  Arms: Pamiparib in combination with Targeted Therapy Drugs

SUMMARY:
The purpose of this study was to investigate the efficacy and safety of pamiparib in patients with EGFR-TKIs-resistant NSCLC, using a single-center, dual-arm, open-label design.

DETAILED DESCRIPTION:
Lung cancer is the second most common cancer type worldwide and remains the leading cause of cancer death worldwide. Non-small cell lung cancer accounts for 80% of the total number of lung cancers, 15-55% of NSCLC have EGFR mutations, of which about 50% of Asians, targeted drugs - epidermal growth factor receptor-tyrosine kinase inhibitors (EGFR-TKIs) ) showed good clinical benefit. However, patients with EGFR-mutant lung cancer experience disease progression within about a year of treatment with EGFR-TKIs, and acquired resistance develops and limits the long-term efficacy of these EGFR-TKIs. About 50% of EGFR-TKIs acquired resistance mutations by the mechanism of T790 mutation. Third-generation EGFR-TKIs can be used to overcome drug resistance against T790 mutation. Unfortunately, acquired resistance to third-generation EGFR-TKIs will eventually emerge, and when third-generation EGFR-TKIs acquire resistance, effective treatment options are still being explored. PARP (poly(ADP-ribose) polymerase) inhibitors represent a new class of anticancer therapy. They exploit synthetic lethality and induce cell death by exploiting defects in DNA repair, poly(ADP-ribose) polymerase-1 (PARP1) and poly(ADP-ribose) polymerase-2 (PARP2) are PARP enzymes Members of the family that play key roles in the DNA damage response (DDR) by acting as DNA damage sensors and signal transducers. PARP inhibitors can be used in combination with conventional NSCLC treatment regimens or as monotherapy. In clinical applications, PARP inhibitors have demonstrated sustained antitumor responses as single agents in BRCA1- or BRCA2-mutated patients. Studies have shown that the single-drug toxicity of PARP inhibitors is much lower than that of platinum drugs, and experimental results in NSCLC cell lines have shown that PARP inhibitors have single-drug activity in NSCLC. The characteristics of the domestic PARP inhibitor, Pamiparib, reflect its advantages over other PARP inhibitors: 1)low drug resistance, 2)high selectivity, 3)high capture of PARP-DNA complexes, 4)high membrane permeability, 5)Dual pathway metabolism, 6)Blood-brain barrier permeability. Multiple clinical data show that Pamiparib as a single agent has favorable safety and antitumor activity in advanced recurrent solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: ≥18 years old
2. Histologically or cytologically confirmed non-small cell lung cancer, and the disease has progressed after first-generation and/or second-generation TKIs treatment with first-line therapy and no T790 mutation, or after third-generation EGFR-TKI treatment After the disease progresses, the guidelines do not recommend a standard protocol.
3. No other concurrent cancer.
4. At least one previously unirradiated lesion that can be accurately measured at baseline with longest diameter ≥ 10 mm (must have a short lymph node excluding axis ≥ 15 mm) according to RECIST criteria with computed tomography (CT), magnetic resonance imaging (MRI) or clinical examination for accurate repeated measures. Or an unevaluable lesion, including but not limited to pleural and ascites, bone metastasis, etc.
5. ECOG physical condition score: 0-3 points.
6. Expected survival period ≥ 3 months.
7. The function of major organs is good, that is, the relevant inspection indicators within 14 days before randomization meet the following requirements: a) Routine blood test:i. Hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); ii. Neutrophil count > 1.5×109/L; iii. Platelet count ≥ 90×109/L; b) Biochemical examination: i. Total bilirubin ≤ 1.5×ULN (upper limit of normal); ii. Blood alanine aminotransferase (ALT) or blood aspartate aminotransferase (AST) ≤ 2.5×ULN; if liver metastasis, ALT or AST ≤ 5×ULN; iii. Endogenous creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); c) Cardiac Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ 50%.
8. Sign the informed consent.
9. The patient is willing and able to comply with the protocol during the study, including receiving treatment and scheduled visits and examinations, including follow-up.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within four weeks.
2. Histologically or cytologically confirmed small cell, large cell neuroendocrine or carcinoid.
3. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as: NYHA class 2 or higher heart failure, unstable angina pectoris, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention of patients.
4. For female subjects: should be surgically sterilized, postmenopausal patients, or agree to use a medically approved contraceptive during the study treatment period and within 6 months after the end of the study treatment period; Serum or urine pregnancy test must be negative within 7 days and must be non-nursing. Male subjects: Patients who should be surgically sterilized, or who agree to use a medically-approved contraceptive method during the study treatment period and within 6 months after the end of the study treatment period.
5. The patient has active pulmonary tuberculosis, bacterial or fungal infection (≥ grade 2 of NCI-CTC, 3rd edition); HIV infection, HBV infection, HCV infection.
6. Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders.
7. The subject has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, thyroid Reduced function; subjects with vitiligo or complete remission of asthma in childhood without any intervention in adulthood can be included; subjects with asthma requiring bronchodilator medical intervention are not included).
8. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 8 weeks
  Total response and partial response ratio

SECONDARY OUTCOMES:
Progression-free survival | 1 year
  Time from randomization to any disease progression and/or death, defined according to strict RECIST (Response Evaluation Criteria in Solid Tumors) v1.1. Lesion will be assessed in comparison to baseline measurements.
Overall survival | 72 weeks
  Randomize time to date of death or last known alive date calculation.
Disease control rate | an average of 1 year
  The proportion of patients with a best response grade of complete response, partial response, or stable disease that has shrunk or stabilized for a period of time.
Objective response rate | 72 weeks
  Assessed according to disease progression as defined by RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
Changes in tumor volume shrinking | 6 months
  Change in tumor volume reduction from randomization to 6 months
Tolerability and Safety | an average of 1 year
  Assessed based on the number of treatment reductions, delays and withdrawals, including the incidence and nature of dose-limiting toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: liu quan, doctor, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The associated efficacy is uncertain.